CLINICAL TRIAL: NCT03750968
Title: Lutein & Zeaxanthin in Pregnancy - Carotenoid Supplementation During Pregnancy: Ocular and Systemic Effects
Acronym: L-ZIP
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Paul S. Bernstein (Other)
Responsible Party: Sponsor-Investigator, Paul S. Bernstein, Professor, Ophthalmology/Visual Sciences, University of Utah
Organization: University of Utah (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: IRB # 116610
Record Dates: First submitted 2018-11-16; First posted 2018-11-23 (Actual); Results first posted 2023-07-11 (Actual); Last update posted 2023-07-11 (Actual); Status verified 2023-06

CONDITIONS: Nutrient Deficiency; Pregnancy Related
MeSH Terms: interventions — Lutein; Zeaxanthins; Control Groups

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Carotenoid group (Experimental): The Carotenoid group will receive a commercially available prenatal vitamin/mineral/Docosahexaenoic acid (DHA) softgel plus a softgel containing lutein/zeaxanthin in safflower oil.
  Interventions: Drug: Carotenoid Group
- Control group (Active Comparator): The Control group will receive the same prenatal vitamin/mineral/Docosahexaenoic acid (DHA) softgel plus a softgel containing only safflower oil.
  Interventions: Dietary Supplement: Control Group

INTERVENTIONS:
Drug: Carotenoid Group — Softgel active ingredients: Lutein 10 mg and Zeaxanthin 2 mg in safflower oil
  Other Names: Softgel with lutein and zeaxanthin
  Arms: Carotenoid group
Dietary Supplement: Control Group — Placebo ingredients: Safflower oil
  Other Names: Softgel without lutein and zeaxanthin
  Arms: Control group

SUMMARY:
This study is designed to test the hypotheses that (1) the third trimester of pregnancy is a period of maternal systemic and ocular carotenoid depletion; (2) prenatal supplementation with 10 milligrams of lutein and 2 milligrams of zeaxanthin will have significant effects on ocular and systemic biomarkers of maternal and infant carotenoid status relative to a matched, standard-of-care prenatal supplement without added lutein and zeaxanthin; and (3) newborn infants with the highest systemic and ocular carotenoid status will have more mature foveal structure.

Mothers will be enrolled in the study during their first trimester, and will take the study carotenoid or control supplements for 6 to 8 months. The final study outcome measurements of mothers and infants will be completed within two weeks of the baby's birth.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women, 18 or older of all races and ethnicities who have an uncomplicated obstetric history and plan to deliver either vaginally or by Caesarian section at the University of Utah for their current pregnancy.

Exclusion Criteria:

* Women who have regularly taken carotenoid supplements containing more than 0.5 mg of lutein and/or zeaxanthin daily during the six months prior to screening
* Women who have significant eye disease associated with macular pigment abnormalities such as Stargardt disease, albinism, or macular telangiectasia type II (MacTel).
* Women with conditions associated with high-risk pregnancy such as adolescent pregnancy, multifetal pregnancy, current or past history of diabetes, pre-eclampsia, previous premature delivery, drug abuse or other significant medical illness

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2019-09-26 (Actual); Primary Completion 2022-01-31 (Actual); Study Completion 2022-01-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul S Bernstein, MD, PhD, Principal Investigator — University of Utah Moran Eye Center
Locations (1):
- University of Utah John A. Moran Eye Center, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Addo EK, Allman SJ, Arunkumar R, Gorka JE, Harrison DY, Varner MW, Bernstein PS. Systemic Effects of Prenatal Carotenoid Supplementation in the Mother and her Child: The Lutein and Zeaxanthin in Pregnancy (L-ZIP) Randomized Trial -Report Number 1. J Nutr. 2023 Aug;153(8):2205-2215. doi: 10.1016/j.tjnut.2023.05.024. Epub 2023 May 27. PMID 37247819
- [Derived] Addo EK, Gorusupudi A, Allman S, Bernstein PS. The Lutein and Zeaxanthin in Pregnancy (L-ZIP) study-carotenoid supplementation during pregnancy: ocular and systemic effects-study protocol for a randomized controlled trial. Trials. 2021 Apr 22;22(1):300. doi: 10.1186/s13063-021-05244-2. PMID 33888136

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Only mothers were considered enrolled. One infant and one mother were considered one unit. The enrollment number and number of participants started/completed represents the number of dyads.
Period: Overall Study
Arm/Group | Carotenoid Group | Control Group
Started | 24 (By definition, only mothers carrying one infant were included in the study. 24 mothers enrolled in the study were assigned to the carotenoid group and out of that, only 21 completed the study. The mother and infant were considered one unit. The 21 mothers and their infants were used for statistical analysis.) | 23 (By definition, only mothers carrying one infant were included in the study. 23 mothers enrolled in the study were assigned to the control group and out of that, only 20 completed the study. The mother and infant were considered one unit. The 20 mothers and their infants were used for statistical analysis.)
Completed | 21 | 20
Not Completed | 3 | 3
Not completed — Adverse Event | 2 | 0
Not completed — Lost to Follow-up | 1 | 3

BASELINE CHARACTERISTICS:
Population: Baseline data were derived from the mothers. Participants who did not complete the final study visit were not included in the analysis.
Groups:
- Carotenoid Group: The Carotenoid group will receive a commercially available prenatal vitamin/mineral/DHA softgel plus a softgel containing lutein/zeaxanthin in safflower oil.
  Carotenoid Group: Softgel active ingredients: Lutein 10 mg and Zeaxanthin 2 mg in safflower oil
- Control Group: The Control group will receive the same prenatal vitamin/mineral/DHA softgel plus a softgel containing only safflower oil.
  Control Group: Placebo ingredients: Safflower oil
- Total: Total of all reporting groups
Arm/Group | Carotenoid Group | Control Group | Total
Number analyzed (Participants) | 21 | 20 | 41
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 21 | 20 | 41
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 30.8 (3.1) | 29.1 (3.7) | 29.9 (1.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 20 | 41
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2
  Not Hispanic or Latino | 20 | 19 | 39
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 21 | 20 | 41
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 21 | 20 | 41
Maternal macular carotenoid levels [Mean (Standard Deviation); unit: unitless] — Macular pigment optical volume is a unitless measure. Details regarding methods and criteria used to assess this outcome measure and interpret the values are in the published protocol available at https://doi.org/10.1186/s13063-021-05244-2 Population: Participants who did not complete a final study visit were excluded from final data analysis.
  unitless | 8809 (3001) | 7002 (2502) | 7906 (2883)
Maternal skin carotenoid levels [Mean (Standard Deviation); unit: Raman units] — Skin carotenoid levels are measured in Raman units. Details regarding methods and criteria used to assess this outcome measure and interpret the values are in the published protocol available at https://doi.org/10.1186/s13063-021-05244-2
  Raman units | 39981 (9495) | 39436 (8733) | 39709 (9021)
Maternal serum carotenoid levels [Mean (Standard Deviation); unit: ng/ml] — We are reporting only lutein + zeaxanthin concentrations. Unit of measurement is nanogram per milliliter (ng/ml).
  ng/ml | 257.6 (116.7) | 217.0 (82.5) | 237.3 (102.3)
Estimated dietary intake of lutein and zeaxanthin [Mean (Standard Deviation); unit: mg/day] — Estimated dietary intake of lutein and zeaxanthin combined is measured in milligrams per day (mg/day). At each study visit, mothers completed the lutein zeaxanthin questionnaire (LZQ™) quantitative food frequency questionnaire that captures ~ 90% of the lutein/zeaxanthin foods consumed in the USA, based on the National Health and Nutrition Examination Survey (NHANES) data.
  mg/day | 4.3 (5.9) | 3.6 (3.1) | 4.0 (4.5)
Smoking habit [Count of Participants; unit: Participants] — Smoking habit is measured on a per participant basis.
  Participants
    Never smoked | 21 | 20 | 41
    Smoked | 0 | 0 | 0
Alcohol intake frequency [Count of Participants; unit: Participants] — Alcohol intake frequency is measured on per participant basis.
  Participants
    Never | 20 | 20 | 40
    Occasional | 1 | 0 | 1
Body mass index (BMI) [Mean (Standard Deviation); unit: kg/m^2] — Unit of measurement is kilogram per meter squared (kg/m^2).
  kg/m^2 | 23.9 (3.7) | 25.4 (4.6) | 24.7 (4.1)

OUTCOME MEASURES:

1. Primary Outcome: Change in Maternal Macular Carotenoid Levels From Enrollment to Birth of Infant
Description: measured in units of macular pigment optical volume (MPOV). Details regarding methods and criteria used to assess this outcome measure and interpret the values are in the published protocol available at https://doi.org/10.1186/s13063-021-05244-2
Time Frame: up to 13 weeks gestation to birth
Population: Participants who did not complete the final study visit were not included in the analysis.
Measure: Mean (Standard Error); unit: unitless
Arm/Group | Carotenoid Group | Control Group
Number analyzed (Participants) | 21 | 20
unitless | 12244 (688) | 7343 (470)

2. Primary Outcome: Change in Maternal Serum Carotenoid Levels From Enrollment to Birth of Infant
Description: We are reporting only lutein + zeaxanthin concentrations. Unit of measurement is in nanograms per milliliter (ng/ml). Details regarding methods and criteria used to assess this outcome measure and interpret the values are in the published protocol available at https://doi.org/10.1186/s13063-021-05244-2
Time Frame: up to 13 weeks gestation to birth
Population: Participants who did not complete the final study visit were not included in the analysis.
Measure: Mean (Standard Error); unit: Nanograms per milliliter
Arm/Group | Carotenoid Group | Control Group
Number analyzed (Participants) | 21 | 20
Nanograms per milliliter | 1030.2 (86.8) | 252.0 (33.4)

3. Primary Outcome: Change in Maternal Skin Carotenoid Levels From Enrollment to Birth of Infant
Description: Maternal skin carotenoid levels are measured in Raman units.
Time Frame: up to 13 weeks gestation to birth
Population: Participants who did not complete a final study visit were excluded from final data analysis.
Measure: Mean (Standard Error); unit: Raman units
Arm/Group | Carotenoid Group | Control Group
Number analyzed (Participants) | 21 | 20
Raman units | 55419 (2421) | 38475 (1932)

4. Secondary Outcome: Infant Macular Carotenoid Levels as Determined by Macular Pigment Optical Density
Description: Comparison of macular carotenoid levels of infants whose mothers received prenatal supplements without carotenoids to those mothers who received prenatal supplements with carotenoids. Details regarding methods and criteria used to assess this outcome measure and interpret the values are in the published protocol available at https://doi.org/10.1186/s13063-021-05244-2
Time Frame: Birth
Population: We report macular pigment optical density for infants whose mothers consented to ophthalmic imaging for their infant.
Measure: Mean (Standard Error); unit: unitless
Arm/Group | Carotenoid Group | Control Group
Number analyzed (Participants) | 12 | 11
unitless | 0.05 (0.01) | 0.04 (0.01)

5. Secondary Outcome: Infant Serum Carotenoid Levels as Determined With High Performance Liquid Chromatography
Description: Comparison of carotenoid levels of infants whose mothers received prenatal supplements without carotenoids to those mothers who received prenatal supplements with carotenoids. We are reporting only lutein + zeaxanthin concentrations. Unit of measurement is nanogram per milliliter (ng/ml). Details regarding methods and criteria used to assess this outcome measure and interpret the values are in the published protocol available at https://doi.org/10.1186/s13063-021-05244-2
Time Frame: Birth
Population: We report data on infants for whom we were able to obtain a blood sample.
Measure: Mean (Standard Error); unit: nanograms per milliliter
Arm/Group | Carotenoid Group | Control Group
Number analyzed (Participants) | 19 | 18
nanograms per milliliter | 270.5 (29.1) | 54.5 (6.6)

6. Secondary Outcome: Infant Skin Carotenoid Levels as Determined With Resonance Raman Spectroscopy
Description: Comparison of carotenoid levels of infants whose mothers received prenatal supplements without carotenoids to those mothers who received prenatal supplements with carotenoids. Infant skin carotenoid levels are measured in Raman units. Details regarding methods and criteria used to assess this outcome measure and interpret the values are in the published protocol available at https://doi.org/10.1186/s13063-021-05244-2
Time Frame: Birth
Population: We report data on infants for whom we were able to obtain skin carotenoid measurements.
Measure: Mean (Standard Error); unit: Raman units
Arm/Group | Carotenoid Group | Control Group
Number analyzed (Participants) | 20 | 20
Raman units | 31656 (1279) | 23011 (869)

ADVERSE EVENTS:
Time Frame: 8 months
Groups:
- Carotenoid Group: The Carotenoid group will receive a commercially available prenatal vitamin/mineral/DHA softgel plus a softgel containing lutein/zeaxanthin in safflower oil. Mother and infant are considered one unit enrolled in the Carotenoid group.
  Carotenoid Group: Softgel active ingredients: Lutein 10 mg and Zeaxanthin 2 mg in safflower oil
- Control Group: The Control group will receive the same prenatal vitamin/mineral/DHA softgel plus a softgel containing only safflower oil. Mother and infant are considered one unit enrolled in the Control group.
  Control Group: Placebo ingredients: Safflower oil
Arm/Group | Carotenoid Group | Control Group
All-Cause Mortality (participants affected / at risk) | 0/24 | 0/23
Serious Adverse Events (participants affected / at risk) | 2/24 | 0/23
Other Adverse Events (participants affected / at risk) | 6/24 | 8/23
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Carotenoid Group (N=24) | Control Group (N=23)
Down syndrome (Congenital, familial and genetic disorders) | 1 (1) | 0 (0) — One infant in the carotenoid group was diagnosed with down syndrome at six weeks of age, which was confirmed by genetic testing. This adverse event originated before study enrollment and was therefore unrelated to the study intervention.
Multiple congenital abnormalities (Congenital, familial and genetic disorders) | 1 (1) | 0 (0) — One infant in the carotenoid group was born prematurely with congenital abnormalities. This adverse event originated before study enrollment and was therefore unrelated to the study intervention.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Carotenoid Group (N=24) | Control Group (N=23)
Gestational diabetes (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 2 (2)
Gestational hypertension (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0)
Pre-eclampsia (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 2 (2)
Anemia (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1)
Exacerbated acne (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0)
Itching (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Torn placenta at delivery (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1)
Cholestasis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Sinus infection (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Worsening depression (Psychiatric disorders) | 1 (1) | 1 (1)
Nose laceration (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
COVID-19 (Infections and infestations) | 2 (2) | 1 (1)
Preterm delivery (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
A limitation of this study was its lack of participant racial, ethnic and socioeconomic diversity. Also, by design, this first-in-humans, randomized clinical trial was limited to low-risk pregnancies. Due to funding and logistical limitations, we could not follow the mothers and their infants beyond their postpartum visit. This meant we were not able to assess the role of maternal breastmilk as a continued source of lutein an zeaxanthin during the first months of life.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-12-21): https://cdn.clinicaltrials.gov/large-docs/68/NCT03750968/Prot_SAP_000.pdf
  • Informed Consent Form (2022-01-12): https://cdn.clinicaltrials.gov/large-docs/68/NCT03750968/ICF_001.pdf